CLINICAL TRIAL: NCT04669717
Title: Pharmacokinetic Considerations and Dosing Strategies of Amoxicillin and Metronidazole or Azithromycin as Adjunct to Non-surgical Periodontal Therapy. A Randomized,6-month, Parallel-group, Clinical Trial.
Brief Title: Antibiotics as Adjuncts to Periodontal Therapy:Pharmacokinetic Considerations and Dosing Strategies
Acronym: AMA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: University of Lausanne (Other)
Responsible Party: Principal Investigator, Catherine Giannopoulou, Professor, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC 2020-01074
Record Dates: First submitted 2020-11-20; First posted 2020-12-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Periodontal Diseases; Antibiotics; Pharmacokinetics
MeSH Terms: conditions — Periodontal Diseases | interventions — Metronidazole

STUDY DESIGN:
Intervention Model Description: Randomized, 3-arm parallel group, single-blind, comparative superiority and exploratory clinical trial with 1:1 allocation ratio.
Who Masked: Investigator
Masking Description: The examiner, the biostatistician and people working in the laboratory for the analyses, will be blinded for the allocation group. Only the two operators and the participants will be aware of the type of treatment based on the computer-generated allocation table that will be kept at the Trial Master File (TMF) of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Amoxicilline and Metronidazole for 7 days (Active Comparator): Drug: AMOXICILLINE Sandoz cpr pell 500mg, Sandoz Pharmaceuticals AG + FLAGYL cpr pell 500mg, Sanofi-Aventis ( Suisse) SA, 3/d for 7 days
  Systemic antibiotics after sub gingival mechanical debridement
  Interventions: Drug: 3/d 500 mg Amoxicilline Sandoz plus 500 mg Flagyl for 7 days
- Amoxicilline and Metronidazole for 3 days (Active Comparator): Drug: AMOXICILLINE Sandoz cpr pell 500mg, Sandoz Pharmaceuticals AG + FLAGYL cpr pell 500mg, Sanofi-Aventis ( Suisse) SA, 3/d for 3 days
  Systemic antibiotics after sub gingival mechanical debridement
  Interventions: Drug: 3/d 500 mg Amoxicilline Sandoz plus 500 mg Flagyl for 3 days
- Azithromycine for 3 days (Active Comparator): Drug: AZITHROMYCIN Pfizer cpr pell 500mg, Pfizer PFE Switzerland GmbH
  1/d 500mg for 3 days
  Systemic antibiotics after sub gingival mechanical debridement
  Interventions: Drug: 1/d 500 mg Azithromycine Pfizer for 3 days

INTERVENTIONS:
Drug: 3/d 500 mg Amoxicilline Sandoz plus 500 mg Flagyl for 7 days — Non-surgical periodontal therapy and radnomly administration of the antibiotics
  Other Names: AMOXICILLINE Sandoz cpr pell 500 mg, Sandoz Pharmaceuticals AG + FLAGYL cpr pell 500 mg, Sanofi-Aventis ( Suisse) SA
  Arms: Amoxicilline and Metronidazole for 7 days
Drug: 3/d 500 mg Amoxicilline Sandoz plus 500 mg Flagyl for 3 days — Non-surgical periodontal therapy and radnomly administration of the antibiotics
  Other Names: AMOXICILLINE Sandoz cpr pell 500 mg, Sandoz Pharmaceuticals AG + FLAGYL cpr pell 500 mg, Sanofi-Aventis ( Suisse) SA
  Arms: Amoxicilline and Metronidazole for 3 days
Drug: 1/d 500 mg Azithromycine Pfizer for 3 days — Non-surgical periodontal therapy and radnomly administration of the antibiotics
  Other Names: AZITHROMYCIN Pfizer cpr pell 500mg, Pfizer PFE Switzerland GmbH
  Arms: Azithromycine for 3 days

SUMMARY:
Periodontitits is a bacteria induced inflammatory disease that destroys the supporting tissues of the tooth and leads to tooth loss. Treatment consists mainly of the mechanical cleaning of the tooth surfaces in order to remove the bacterial deposits (plaque and calculus). This procedure can reduce the level of pathogenic bacteria but it can not eradicate them. In severe cases, for the complete resolution of the disease, the elimantion of certain species of bacteria is needed. In order to achieve that, the combination of different regimens of antibiotics adjunctive to the mechanical treatment has been proposed. However, dosage and duration of antimicrobial therapy should be optimal and not excessive as issues may arise related to increased antimicrobial resistance in the population and the individual due to habitual prescription of wide-spectrum antibiotic regimens, horizontal gene transfer and genetic mutation.

In the present study, in an effort to optimize the dosage and duration of the antimicrobial regimen, we will determine the pharmacokinetics (PK) and pharmacodynamic (PD) properties of the MET-AMO combination and of AZI in Gingival Crevicular Fluid (GCF), saliva and serum in severe periodontitis patients during and after either a 3-day or a 7-day course of treatment.

DETAILED DESCRIPTION:
This is a randomized, 3-arm parallel group, single-blind, comparative superiority and exploratory clinical trial of 44 months involving 45 patients with periodontitis attending the Division of Regenarative Dental Medecine and Periodontology of the University of Geneva. First, a routine clinical and radiographic periodontal examination will be conducted by a periodontist. Treatment will be done in 2 appointments by mechanical debridement of the diseased sites by two experienced clinicians. At the end of the treatment, one third of the patients will be assigned for treatment with 500mgAMO+ 500mgMET 3 times a day during 1 week, one third for treatment with 500mgAMO+ 500mgMET 3 times a day during 3 days and the last third for treatment with 500mg AZI once a day for 3 days.

Clinical samples will be taken at Days 0, 2, 4 and 8 after the start of the antibiotic administration . Gingival Crevicular Fluid (GCF) will be collected from four sites with paperpoints, blood sample by finger puncture, unstimulated saliva and subgingival plaque from four sites with paper points. The concentration and duration effect of AMO+MET and AZI in GCF, saliva and serum will be assessed in the Laboratory of Clinical Pharmacology at the University Hospital of Lausanne (CHUV) by high performance liquid chromatography coupled to tandem mass spectrometry (LC-MS/MS). The microbiological effect on 6 selected organisms will be assessed by RT-PCR at 3 and 6 months after treatment. The clinical results will be evaluated 6 months later. The study duration for the patient will be approximately 8 months.

All adverse events (AE) and all serious adverse events (SAEs) will be recorded and addressed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Aged 18-80 years old with need of periodontal treatment associated with adjunctive antibiotic therapy
* Presence of at least 30% of the teeth in the mouth with PD>6mm and BOP

Exclusion Criteria:

* Persons with systemic illnesses (uncontrolled diabetes mellitus, cancer, human immunodeficiency virus, bone metabolic diseases or disorders that compromise wound healing, radiation, or immunosuppressive therapy)
* Pregnancy or lactation
* Persons who had taken AB within the previous 2 months
* Persons who are taking nonsteroidal anti-inflammatory drugs
* Persons who have a confirmed or suspected intolerance to 5-nitroimidazole derivatives or amoxicillin or macrolides
* Previous periodontal therapy the last 1 year
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow due to language problems, psychological disorders, dementia, etc. of the participant
* Participants not willing to attend regular dental maintenance visits and follow-up evaluations
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The concentration of AMO+MET and AZI in GCF, saliva and serum | At Day 0,2,4,8 post-dose
  The concentration of the drugs will be assessed in samples of gingival crevicular fluid, saliva and serum at days 0, 2, 4 and 8 after the start of the antibiotic administration.The concentration of the studied antibiotics in the different fluids will be expressed as ng/ml

SECONDARY OUTCOMES:
Differences between the three treatment arms in the proportion of participants classed as treatment success at 6 months; defined as absence of sites with PD ≥ 5 mm and concomitant bleeding on probing. | At Month 3 and Month 6 post-intervention
  Comparisons between groups assessed at 3 and 6 months after treatment
Differences between the three treatment arms in the levels of 6 organisms in subgingival plaque samples. For those bacteria with a threshold of >1000cells/ml, results will be expressed as median counts. | At Month 3 and Month 6 post-intervention
  Comparisons between groups will be assessed at 3 and 6 months after treatment
Number of participant per treatment arm with adverse events as a mesure of safety. | At Day 2, Day 4 and Day 8 post-intervention
  Adverse events will be collected from the start of study treatment and until the end of the study (at 6 months evaluation)
Patient's compliance will be evaluated | At Day 8 after intervention
  Compliance will be evaluated by pill count at the end of the antibiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Giannopoulou, Dr med dent, Principal Investigator — University Clinics of Dental Medicine, University of Geneva
Locations (1):
- University of Geneva, University Clinics of Dental Medicine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giannopoulou C, Cionca N, Almaghlouth A, Cancela J, Courvoisier DS, Mombelli A. Systemic Biomarkers in 2-Phase Antibiotic Periodontal Treatment: A Randomized Clinical Trial. J Dent Res. 2016 Mar;95(3):349-55. doi: 10.1177/0022034515618949. Epub 2015 Nov 24. PMID 26604272